CLINICAL TRIAL: NCT04182503
Title: Investigation on the Health Effects of Environmental and Behavioral Factors on Embryonic Development and Pregnancy Based on Internal and External Exposure Monitoring
Brief Title: Environmental Factors and Embryonic Development Project
Acronym: EFED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Collaborators: Peking University (Other); Sun Yat-sen University (Other); Shandong University (Other); Zunyi Medical College (Other); Zhejiang University (Other); Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, SHANG Xue-jun, Professor, Jinling Hospital, China
Other Study IDs: 2018YFC1004300
Record Dates: First submitted 2019-11-12; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Spontaneous Abortion; Fetal Death; Stillbirth; Birth Defects; Preterm Birth; Low Birth Weight; Pregnancy With Medical Condition (Non-Specific); Gestational Diabetes; Gestational Hypertension
MeSH Terms: conditions — Abortion, Spontaneous; Fetal Death; Stillbirth; Congenital Abnormalities; Premature Birth; Diabetes, Gestational; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators will collect a 8 ml blood sample and a 10 ml urine sample from each pregnant woman at their first pregnancy examination, and a 10 ml cord blood sample at delivery. The blood sample will be separated into plasma/serum and white blood cells/blood clots shortly after collection and then stored at -80 degrees celsius. The urine sample will be separated into several tubes before storage at -80 degrees celsius.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (16):
- Beijing
  Interventions: Other: No intervention
- Guangzhou
  Interventions: Other: No intervention
- Jinan
  Interventions: Other: No intervention
- Nanjing
  Interventions: Other: No intervention
- Hangzhou
  Interventions: Other: No intervention
- Wuhan
  Interventions: Other: No intervention
- Zunyi
  Interventions: Other: No intervention
- Xiangyang
  Interventions: Other: No intervention
- Nantong
  Interventions: Other: No intervention
- Suizhou
  Interventions: Other: No intervention
- Huangshi
  Interventions: Other: No intervention
- Changzhou
  Interventions: Other: No intervention
- Suqian
  Interventions: Other: No intervention
- Shiyan
  Interventions: Other: No intervention
- Xiaogan
  Interventions: Other: No intervention
- Huanggang
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a multi-city observational cohort study without intervention.

SUMMARY:
The Environmental Factors and Embryonic Development Project was set up to investigate environmental exposures and behavioral factors responsible for embryonic dysplasia and gestational complications in pregnant women.

DETAILED DESCRIPTION:
The Environmental Factors and Embryonic Development Project is about to recruit pregnant women from 16 cities, including Beijing, Guangzhou, Jinan, Nanjing, Hangzhou, Wuhan, Zunyi, Xiangyang, Nantong, Suizhou, Huangshi, Changzhou, Suqian, Shiyan, Xiaogan, and Huanggang. The project plans to recruit 6000-12000 participants in each city. Biological samples, questionnaires and data for embryonic dysplasia and gestational complications of pregnant women will be collected. The study includes four stages. In the first stage, the investigators will identify external environmental factors and behavioral factors that are associated with embryonic dysplasia and gestational complications in pregnant women based on external exposure monitoring strategies. In the second and third stages, the investigators will conduct several nested case-control studies based on our prospective cohort. Internal exposure monitoring will be applied to identify environmental endocrine disruptors which are associated with embryonic dysplasia and gestational complications in pregnant women in the second stage. In the third stage, the investigators will conduct genome-wide association study (GWAS) to screen susceptible genes or polymorphisms that are associated with embryonic dysplasia and gestational complications in pregnant women, identify any gene-environmental interactions with reference to the findings of the 1st and 2nd stages, and finally establish a comprehensive disease risk prediction model. In the fourth stage, the investigators will build animal models in order to identify the mechanisms how high-risk environmental exposures or behavioral factors as identified in the above stages may lead to embryonic dysplasia and gestational complications in pregnant women. The research team of the 16 cities are from Peking University (Beijing), Sun Yat-sen University (Guangzhou), Shandong University (Jinan), Chinese People's Liberation Army Eastern Theater General Hospital (Nanjing, Nantong, Changzhou, and Suqian), Zhejiang University (Hangzhou), Huazhong University of Science and Technology (Wuhan, Xiangyang, Suizhou, Huangshi, Shiyan, Xiaogan, and Huanggang), Zunyi Medical University (Zunyi), respectively. The core members of each research team are composed of experts from different disciplines in the field of public health.

ELIGIBILITY:
Inclusion Criteria:

1. pregnancy within 13 weeks;
2. age between 20-45 years;
3. natural conception;
4. singleton pregnancy;
5. living in the local area for one year or more.

Exclusion Criteria:

1. pregnant women with serious chronic diseases and infectious diseases (such as cancer, chronic cardiovascular and cerebrovascular diseases, chronic renal failure, HIV infection);
2. have participated in other scientific research projects;
3. refuse to participate or are unwilling to sign informed consent.;
4. are unable to guarantee delivery in our designated hospitals.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women attending their first routine antenatal examinations.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of spontaneous abortion | up to 28 gestational weeks
Incidence of fetal death/stillbirth | after 20 gestational weeks to delivery
Incidence of birth defects | Delivery
Incidence of low birth weight | Delivery
Incidence of preterm birth | Delivery
Incidence of pregnancy with heart disease | During pregnancy (up to 10 months)
Incidence of pregnancy with hyperthyroidism | During pregnancy (up to 10 months)
Incidence of gestational diabetes | During pregnancy (up to 10 months)
Incidence of gestational hypertension | During pregnancy (up to 10 months)

CONTACTS AND LOCATIONS:
Overall Officials: Xuejun Shang, PhD, Principal Investigator — Jinling Hospital, China
Locations (19):
- China (19):
  - Haidian Maternal and Child Healthcare Hospital, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Meitan People's Hospital, Zunyi, Guizhou
  - Renhuai Hospital of Traditional Chinese Medicine, Zunyi, Guizhou
  - The First Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The Second Affliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - People's Hospital of Qichun County, Huanggang, Hubei
  - Huangshi Maternal and Child Healthcare Hospital, Huangshi, Hubei
  - Shiyan Maternal and Child Healthcare Hospital, Shiyan, Hubei
  - Maternal and Child Healthcare and Family Planning Service Center of Zengdu District, Suizhou, Hubei
  - Huangpi Maternal and Child Healthcare Hospital, Wuhan, Hubei
  - Maternal and Child Healthcare Hospital of HuBei, Wuhan, Hubei
  - Xiangyang No. 1 People's Hospital, Hubei University of Medicine, Xiangyang, Hubei
  - Anlu Maternal and Child healthcare Hospital, Xiaogan, Hubei
  - Changzhou Second People's Hospital, Changzhou, Jiangsu
  - Nantong Maternal and Child Healthcare Hospital, Nantong, Jiangsu
  - Shuyang Hospital Affiliated to Xuzhou Medical University, Suqian, Jiangsu
  - Center for Reproductive Medicine, Shandong University, Jinan, Shandong
  - Women's Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided